CLINICAL TRIAL: NCT07269587
Title: A Retrospective, Observational, and Multicenter Real-world Study on the Treatment of Adult B-cell Acute Lymphoblastic Leukemia With CNCT-19
Brief Title: A Real-world Study on the Treatment of Adult B-cell Acute Lymphoblastic Leukemia With CNCT-19
Status: Active, not recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jin Wang, chief physician, MD, PhD, Ruijin Hospital
Other Study IDs: CN-ALL RWS001
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: ALL (Acute B-Lymphoblastic Leukemia); CAR-T Cell Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observation group
  Interventions: Drug: CNCT-19

INTERVENTIONS:
Drug: CNCT-19 — All patients have received CNCT-19

SUMMARY:
This clinical study is a retrospective, observational, and multicenter post marketing real-world study aimed at evaluating the efficacy and safety of CNCT-19 in the treatment of Chinese adult B-cell acute lymphoblastic leukemia patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 14 years old;
2. Diagnosed with CD19+B-cell acute lymphoblastic leukemia [refer to the Chinese Guidelines for Diagnosis and Treatment of Adult Acute lymphoblastic Leukemia (2024 edition)];
3. Patients who have received treatment with CNCT-19.

Exclusion Criteria:

1. Individuals with acute graft-versus-host disease (GVHD) or moderate to severe chronic GVHD within the first 4 weeks of screening; Individuals who have received systemic drug therapy for GVHD within the past 4 weeks prior to reinfusion;
2. Active systemic autoimmune diseases during treatment;
3. Those who meet any of the following criteria:

   * Positive hepatitis B surface antigen (HBsAg) and/or hepatitis B e antigen (HBeAg);
   * hepatitis B e antibody (HBe Ab) and/or hepatitis B core antibody (HBc Ab) are positive, and the number of HBV-DNA copies is greater than the measurable lower limit;
   * Hepatitis C antibody (HCV Ab) positive;
   * Positive for Treponema pallidum antibody (TP Ab);
   * Positive human immunodeficiency virus (HIV) antibody test;
   * EBV-DNA and CMV-DNA copy numbers are greater than the measurable lower limit;
4. Individuals known to have a history of hypersensitivity reactions to the components of the formulation used in the experiment.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients received CNCT-19 treatment in all participant center of this study
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2025-11-07 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
overall response rate(for R/R patients) | Till the end of the study, up to 24 months
  The proportion of patients who reach CR/CRi.Bone marrow of every patient will be analysed by multiparameter flow cytometry or/and RT-qPCR for MRD evaluation.
minimal residual disease negativity rate(for MRD positive patients) | Till the end of the study, up to 24 months
  The proportion of patients who reach MRD negative in all patients reached CR/CRi.Bone marrow of every patient will be analysed by multiparameter flow cytometry or/and RT-qPCR for MRD evaluation.

SECONDARY OUTCOMES:
DOR(Duration Of Remission) | till the end of the study, up to 24 months
  Time from the first assessment of MRD negative to the first assessment of MRD positive or death from any cause.
rate of Allogeneic hematopoietic stem cell transplantation | till the end of the study, up to 24 months
  The proportion of patients who receive allo-HSCT after CNCT19 treatment.
Relapse-free survival (RFS) | till the end of the study, up to 24 months
  Interval from the date of treatment of the CNCT-19 to the time of hematological recurrence or death from any cause. Evaluation of RFS will be based on follow-up results.
Overall Survival(OS) | till the end of the study, up to 24 months
  Interval from the date of the feedback to the time of death due to any reason. Evaluation of OS will be based on follow-up results.
incidence of Adverse Events(AEs) | up to 24 months
  The proportion of patients who have adverse events after CNCT-19 treatment.Adverse events will be assessed by CTCAE v5.0
incidence of Severe Adverse Events(SAEs) | up to 24 months
  The proportion of patients who have severe adverse events after CNCT-19 treatment.Adverse events with one of the following damages should be classified as serious drug adverse events:
  1. Causing death;
  2. Endangering life;
  3. Causing hospitalization or prolonged hospitalization time;
  4. Causing permanent or significant disability/loss of function;
  5. Congenital abnormalities/birth defects;
  6. Causing other important medical events that, if left untreated, may result in the situations listed above.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided